CLINICAL TRIAL: NCT06862687
Title: The Effect of Cold Application Using Two Different Methods on Arteriovenous Fistula Pain
Brief Title: Arteriovenous Fistula Pain and Cold Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehtap KAVURMACI, Prof, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B.30.2.ATA.0.01.00/300
Record Dates: First submitted 2025-02-27; First posted 2025-03-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Arteriovenous Fistula Pain
Keywords: Arteriovenous Fistula; cold application; Hemodialysis; Kidney Failure; Pain
MeSH Terms: conditions — Arteriovenous Fistula; Renal Insufficiency; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Group Assignment (Active Comparator): Three different interventions (cooling spray, aloe vera gel, and standard procedure) were applied to participants in sequence
  Interventions: Other: Cooling Spray; Other: Cold Aloe Vera Gel Application; Other: Standard Procedure (Control Condition)

INTERVENTIONS:
Other: Cooling Spray — A cooling spray containing propan-butane-pentane was applied 25 cm from the cannulation site until mild whitening/frosting appeared.
  The standard AVF cannulation procedure was performed. Pain levels were measured immediately after the procedure using VAS.
Other: Cold Aloe Vera Gel Application — 1 ml of cold aloe vera gel was applied to a 5x5 cm area over the fistula site. The standard AVF cannulation procedure was conducted. Pain levels were assessed post-procedure using VAS.
Other: Standard Procedure (Control Condition) — No additional pain-relief intervention was applied. The nurse performed the standard AVF cannulation procedure, including hand hygiene, thrill assessment, and site disinfection.
  Pain levels were assessed immediately after cannulation using the Visual Analog Scale (VAS).

SUMMARY:
TThis study was designed as a single-group comparative prospective intervention study. The aim of the study was to assess the effectiveness of different pain management interventions during AVF cannulation. The effects of pain management methods such as cooling spray, aloe vera gel, and the standard procedure on pain levels, and which intervention was more effective in reducing pain compared to the standard procedure, were investigated.

The study included patients over 18 and under 65 years old, undergoing hemodialysis, having an AVF, literate, without an aloe vera allergy, and without communication barriers or psychiatric disorders.

The main research questions were defined as follows: Did different pain management methods (cooling spray, aloe vera gel, and standard procedure) affect pain levels during AVF cannulation? Which intervention was more effective in reducing pain levels? The primary hypotheses were defined as The application of cooling spray and aloe vera gel would reduce pain levels more than the standard procedure.

The researchers compared pain levels after each intervention to determine which one was more effective. Three different interventions (cooling spray, aloe vera gel, and standard procedure) were applied to participants in sequence, and pain levels were assessed after each intervention using the Visual Analog Scale (VAS). Additionally, feedback from participants regarding each intervention was collected.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 and under 65 years old
* Literate
* Have an arteriovenous fistula (AVF)
* Undergoing hemodialysis (HD) treatment at least twice a week
* No allergy to aloe vera
* No communication barriers and/or psychiatric disorders

Exclusion Criteria:

* Diagnosed with malignancy
* Having any sensory problems that prevent the assessment of perception and pain
* Using any analgesic preparations
* Having a vascular access other than AVF
* Patients in whom AVF cannulation is not successful in a single attempt

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Pain Level (VAS - Visual Analog Scale) | 3 months
  The pain level experienced by patients after AVF cannulation was assessed using the VAS (0-10 scale).
  Pain scores were recorded and compared across all three interventions. Lower VAS scores indicate greater effectiveness of the intervention in pain reduction. n this scale, patients are asked to describe their pain using numbers, where "0" represents no pain and "10" indicates the highest, unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Research Hospital, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thompson J, Steinheiser MM, Hotchkiss JB, Davis J, DeVries M, Frate K, Helm R, Jungkans CW, Kakani S, Lau S, Lindell K, Landrum KM, McQuillan KA, Shannon DJ, Wuerz L, Pitts S. Standards of care for peripheral intravenous catheters: evidence-based expert consensus. Br J Nurs. 2024 Nov 21;33(21):S32-S46. doi: 10.12968/bjon.2024.0422. PMID 39585227